CLINICAL TRIAL: NCT06662526
Title: Trace Lithium Dosage for Prevention of Cognitive Declining in Patients with Mood Illnesses: a Randomized Double Blind Placebo Controlled Trial
Brief Title: Lithium for Prevention of Cognitive Declining in Mood Illnesses
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Paul Vohringer, Associate profesor of psychiatry, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 002085
Record Dates: First submitted 2024-09-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Dementia; Bipolar Disorder (BD); Depression - Major Depressive Disorder; Mild Cognitive Impairment (MCI)
Keywords: Lithium trace doses; mood disorders; cognitive declining prevention; dementia prevention
MeSH Terms: conditions — Dementia; Bipolar Disorder; Cognitive Dysfunction; Mood Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trace lithium dose (Experimental): This arm will consist of 125 participants, each receiving trace doses of lithium
  Interventions: Drug: Trace lithium dose plus treatment as usual
- Placebo (Placebo Comparator): This arm will consist of 125 participants, each receiving placebo.
  Interventions: Drug: Placebo pill plus treatment as usual

INTERVENTIONS:
Drug: Trace lithium dose plus treatment as usual — Subjects assigned to the active arm will receive 50 mg of lithium per day, for five years
  Arms: Trace lithium dose
Drug: Placebo pill plus treatment as usual — Patients will receive a placebo pill plus treatment as usual by their clinical providers
  Arms: Placebo

SUMMARY:
INTRODUCTION: Mood disorders, bipolar disorder and recurrent unipolar depression, are among the most common mental health conditions worldwide. Patients with mood conditions are considered a high-risk group for cognitive impairment. Specifically, the risk estimates for developing dementia range from 1.90 to 3.02 for MDD, and 2.36 to 5.58 for mood conditions. Mild cognitive impairment (MCI), is an intermediate stage between the expected cognitive decline of normal aging and the more serious decline of dementia. On the other hand, Lithium has long been recognized as the gold standard treatment for mood conditions and the eventual effect as neurocognitive agent. It has been reported that long-term treatment with lithium decreased the prevalence of dementia compared to patients not receiving lithium treatment. The prevalence of Alzheimer is lower in patients with bipolar disorder who are on chronic lithium therapy compared to those who are not, and low-dose lithium (from 300 mcgr to 50 mg/day) may provide neuroprotective benefits without significant side effects. This trace dosage is hypothesized to be sufficient to activate neuroprotective pathways while minimizing toxicity.

AIM: to investigate the effect of trace dosage of lithium on cognitive function in individuals at risk of developing these conditions. Specifically, this study will randomize healthy participants and patients with mild cognitive impairment to receive either a low-dose lithium supplement (50 mg daily) or a placebo, with the primary outcome being the incidence of MCI or worsening of the preexisting MCI.

HYPOTHESIS: Patients with mood conditions exposed to trace lithium dosage will have a smaller incidence of MCI or less worsening of the preexisting MCI compared with patients receiving placebo.

GOALS: A)To examine the effectiveness of lithium in prevention of mild cognitive impairment in patients with the high-risk factor of preexisting mood illnesses (i.e., unipolar depression or bipolar illness). The primary outcome is incidence of newly diagnosed mild cognitive impairment (MCI) or worsening of preexisting MCI. B) To assess, in an exploratory analysis, the clinical predictors of good lithium response in this sample. These analyses will also assess lithium effects on suicide, mortality, quality of life, functional impairment, and overall medical morbidity.

METHODOLOGY: The study will be double-blind randomized placebo-controlled trial. Patients will be recruited from two sites in Santiago, Chile, the Psychiatric Institute Dr. José Horwitz Barak and the Psychiatric Clinic of the University of Chile. Subjects aged 55 to 75 years, who present mood disorders and are not currently on lithium therapy, will be invited to participate. Inclusion Criteria are: Age 55-75, DSM-5 diagnosis of major depressive disorder or bipolar disorder (types I or II), current or lifetime, prior to participation in this study, each subject must sign an informed consent. Exclusion Criteria are: current mood treatment with lithium, alcohol dependency within the past month, current serious unstable medical conditions or history of medical illness that would contraindicate a trial of lithium, current or past severe kidney disease or baseline creatinine higher than 1.5 mg/dl, active suicidal ideation with plan and intent (Columbia Suicide Severity Rating Scale Screen Version (C-SSRS Screen) higher than points), current or past severe thyroid disease or baseline TSH higher than 5.0 uUI/dl, current diagnosis of dementia of any kind. Participants will be randomized into one of two arms: a trace dose lithium or placebo, each group consisting of 125 subjects. Block randomization will be stratified by diagnosis (bipolar vs MDD), gender, decade of age, and presence or absence of any baseline cognitive impairment Interventions. All participants will receive their usual clinical medical treatment during the time the study is conducted. All psychotropic medications will be allowed to be given per standard of care except lithium. The study defined randomization to lithium or placebo arms as adjuncts to other medications. Intervention arm will consist in lithium 50 mg oral tablets per day (trace doses). Control arm will consist in placebo tablet.

OUTCOME: The primary outcome measure will be the incidence of Mild Cognitive Impairment (MCI) or worsening of preexisting MCI at one, three, and four years. This primary outcome will be defined as change from patients initially with a Clinical Dementia Rating Scale (CDR) score of 0 to 0.5 (MCI) or patients initially with a score in the CDR of 0.5 that change to 1. (worsening of MCI). The primary analysis will employ a Cox regression model to analyze the time to first clinical diagnosis of MCI or worsening of MCI.

DETAILED DESCRIPTION:
Mood disorders, bipolar disorder and recurrent unipolar depression, are among the most common mental health conditions worldwide. Research estimates that the international lifetime prevalence of bipolar disorder (BD) is 0.8% for Type 1 and up to 2% for Type 2 while for major depressive disorder (MDD), prevalence rates stand between 6.4%. Additionally, in Chile lifetime prevalence for MMD is 9.2% and 2% for any bipolar disorder.

It has been extensively suggested by research that patients with mood conditions are considered a high risk group for cognitive impairment. Among those, mild cognitive impairment (MCI), is an intermediate stage between the expected cognitive decline of normal aging and the more serious decline of dementia. It is considered a transitional-preclinical stage between healthy aging and dementia. Over time, various definitions have been proposed for MCI and its subtypes, but in general, it is characterized by a measurable decline in one or more cognitive domains, such as memory, attention, language, executive function, or visual skills, that exceeds what might be expected based on an individual's age and education background, but does not markedly impair the individual's independence in everyday activities; it is also characterized by concerns about these cognitive changes, either reported by the patient or an informant. While not all individuals with mild MCI will go on to develop dementia, evidence suggests that those with this condition are at a higher risk, with annual conversion rates ranging from 8% to 15% per year. This is why detecting and treating MCI represents a critical opportunity for early intervention and potentially preventing or delaying the onset of more severe neurodegenerative diseases. Dementia is a general term to describe a condition characterized for a group cognitive and behavioral symptoms, observed in several conditions. According to the National Institute on Aging-Alzheimer's Association, it can be defined as the decline from previous levels of functioning and performing in at least two of the following areas, that must interfere with the usual functioning: 1) the ability to acquire and remember new information, 2) reasoning and handling of complex tasks or poor judgment, 3) visuospatial abilities, 4) language functions and 5) personality, behavior, or comportment. Among all causes of dementia, Alzheimer Disease (AD) is the most common form, representing 60-70% of cases.

There is substantial body evidence indicating that major MDD and BD are closely linked to the development of mild cognitive impairment (MCI) and dementia. Research has shown that individuals with affective disorders are particularly vulnerable, exhibiting a markedly higher risk of developing dementia and other neurodegenerative conditions, compared to the general population. Specifically, the risk estimates for developing dementia range from 1.90 to 3.02 for MDD, and 2.36 to 5.58 for BD. Further, people suffering affective disorders have also a 2.5 times higher risk of developing dementia when compared to other medical conditions like osteoarthritis of diabetes. This increased risk is thought to be associated with factors such as the chronic nature of bipolar disorder, the impact of mood episodes on cognitive function, and the potential shared underlying pathophysiological mechanisms between the two conditions.

Another important clinical aspect with this high risk of MCI and dementia group is pertained with earlier presentation of cases when compared with the general population. The pathophysiology underlying cognitive decline in mood disorders involves neuroinflammation, oxidative stress, mitochondrial dysfunction, and impaired neuroplasticity, all of which overlap with mechanisms observed in neurodegenerative conditions such as MCI and Alzheimer's disease (AD).

Lithium Evidence as Cognitive Protector Agent Lithium has long been recognized as the gold standard treatment for bipolar disorder, and has also played a significant role as an adjunct therapy for major depressive disorder. In recent years, however, the scientific community has shown increasing interest in the potential therapeutic applications of lithium beyond its traditional use in the management of BD and MDD. One particularly promising area is the prevention of cognitive decline in affective disorders. A growing body of evidence has suggested that lithium may possess neuroprotective properties, which could be leveraged to address the pressing challenges of dementia, MCI and other neurodegenerative disorders like Parkinson disease among others.

Research conducted to determine the underlying mechanisms of the potential neuroprotective effects of lithium have shown a diversity of targets. Its neuroprotective potential may be attributed to its ability to modulate several key cellular pathways involved in the pathogenesis of neurodegenerative disorders. For instance, lithium has been shown to inhibit glycogen synthase kinase-3 (GSK-3), a kinase that plays a central role in the hyperphosphorylation of tau protein, a hallmark pathological feature of Alzheimer's disease. This inhibition of GSK-3 by lithium helps to reduce the accumulation of hyperphosphorylated tau, which is a major contributor to the formation of neurofibrillary tangles, one of the characteristic hallmarks of Alzheimer's disease pathology. Moreover, lithium has also been found to enhance the activity of brain-derived neurotrophic factor (BDNF), a crucial neurotrophin involved in neuronal survival, synaptic plasticity, and neurogenesis - all of which are compromised in the context of neurodegenerative diseases. The increased availability of BDNF due to lithium treatment has been shown to promote neuronal health and resilience, thereby mitigating the progression of neurodegenerative processes. Additionally, lithium exerts anti-inflammatory and antioxidant effects, which have been linked to its neuroprotective properties. Moreover, it may also exert its neuroprotective effects by inducing increases in the levels of the anti-apoptotic factor Bcl-2, thereby suppressing neuronal death and promoting cell survival. This action of lithium to enhance Bcl-2 levels and inhibit apoptosis has been observed in various in vitro and in vivo models of neurodegenerative conditions, suggesting that it is a key mechanism through which lithium produces its neuroprotective properties. Additionally, lithium has been found to modulate oxidative stress pathways, mitochondrial function, and neuroinflammation - all of which are implicated in the etiology of neurodegenerative disorders. By targeting these multiple pathways, lithium exhibits a multifaceted approach to neuroprotection, which may contribute to its potential therapeutic utility in the prevention and management of dementia and related neurodegenerative conditions. Taken together, these findings suggest that lithium may hold significant promise as a therapeutic agent for the prevention and management of dementia and other neurodegenerative conditions.

Neurocognitive role of lithium the prevention of dementia in affective disorders.

Seminal clinical evidence coming from a cohort of patients with mood illnesses followed for more than twenty years was reported in 2007. It was observed that long-term treatment with lithium in these subjects was associated with lower prevalence of dementia compared to patients not receiving lithium treatment . Other case-control study found that the prevalence of Alzheimer's disease was significantly lower in elderly euthymic patients with bipolar disorder who were on chronic lithium therapy compared to those who were not.

One promising avenue of research is the use of lithium in preventing mild cognitive impairment (MCI) and dementia. Recent research suggests that low-dose lithium (from 300 mcgr to 50 mg/day) may provide neuroprotective benefits without significant side effects. This trace dosage is hypothesized to be sufficient to activate neuroprotective pathways while minimizing toxicity.

This proposal aims to investigate the effect of lithium on cognitive function in individuals at risk of developing these conditions. It is intended to determine the potential benefits of lithium in mitigating the progression of cognitive decline. Additionally, this research will contribute to our understanding of the role of lithium in neuroprotection and its potential implications for public health interventions aimed at reducing the burden of neurodegenerative disorders.

The present study aims to build upon this existing evidence by examining the efficacy of lithium trace supplementation in preventing cognitive decline and dementia in a large, well-designed randomized controlled trial. Specifically, this study will randomize cognitively healthy patients with mood disorders or patients with preexisting MCI to receive either a low-dose lithium supplement (50 mg daily) or a placebo, with the primary outcome being the incidence MCI or worsening of the preexisting MCI

II. HYPOTHESIS General Patients with mood conditions exposed to trace lithium dosage will have a smaller incidence of MCI or less worsening of preexisting MCI compared with patients receiving placebo.

Specific A. Trace dosage of lithium (50 mg/day) will be efficacious in preventing newly diagnosed MCI or worsening in existing MCI, in patients with mood conditions compared with patients receiving placebo.

B. There will not be a differential rate of adverse events related to trace lithium dosage compared with placebo.

C. There will be clinical features that may predict the lithium response in the active arm.

III. GOALS

General Goals:

A. To examine the effectiveness of lithium in prevention of mild cognitive impairment in patients with the high-risk factor of preexisting mood illnesses (i.e., unipolar depression or bipolar illness). The primary outcome is incidence of newly diagnosed mild cognitive impairment (MCI) or worsening of preexisting MCI.

B. To assess, in an exploratory analysis, the clinical predictors of good lithium response in this sample. These analyses will also assess lithium effects on suicide, mortality, quality of life, functional impairment, and overall medical morbidity.

Specific Goals:

For General Goal A

1. Determine the incidence rate of newly diagnosed MCI in the lithium and placebo groups.
2. Determine the incidence of worsening of already diagnosed MCI in the lithium and placebo groups
3. Compare the cognitive decline trajectories in time for both groups.
4. Measure cognitive function using standardized assessments over the study period.
5. Compare the progression of profiles of cognitive decline between the two groups.

For General Goal B:

1. Identify demographic and clinical predictors of a positive response to lithium.
2. Assess the impact of lithium on secondary outcomes like quality of life and functional impairment.
3. Monitor and document any adverse events associated with lithium treatment
4. Analyze the safety profile of trace lithium dosage.

Procedures In each of the mentioned psychiatric facilities, eligible subjects will be invited to participate in the study as part of their primary care psychiatry. In case of interest, they will be contacted by one of the study's researchers to confirm that the eligibility criteria are met. Those subjects who meet the inclusion criteria and do not meet the exclusion criteria at baseline assessment will be included in the trial. After giving consent, subjects will be invited to undergo the baseline assessment.

Randomization Participants will be randomized into one of two arms: a trace dose lithium or placebo, each group consisting of 125 subjects. Block randomization will be stratified by diagnosis (bipolar vs MDD), gender, decade of age, and presence or absence of any baseline cognitive impairment (defined clinically as the presence of executive dysfunction, attentional impairments, and/or poor working or short-term memory). Equipoise randomization, as has been implemented in other RCTs, will be used to minimize risks by allowing subjects and/or clinicians to exclude one of the two treatment arms if past clinical history and/or patient preferences indicate an undue risk for side effects in one of the arms.

Interventions All participants will receive their usual clinical medical treatment during the time the study is conducted. All psychotropic medications will be allowed to be given per standard of care except lithium. The study defined randomization to lithium or placebo arms as adjuncts to other medications.

* Intervention arm: Lithium 50 mg oral tablets per day (trace doses).
* Control arm: placebo tablet.

Assessments In both groups, the assessments will be carried out at the baseline and subsequently every six months over the next four years by blind researchers. Research study investigators will base this diagnosis on interviews with the patient, caregivers, clinicians, and/or chart assessments.

Data Analysis The primary analysis (by full intention-to-treat) will be a survival analysis of time to either detection of MCI or worsening of MCI as defined for the primary outcome during the scheduled treatment period of patients allocated to lithium versus placebo. Time to first event (newly diagnosed MCI or worsening of an already existing one) during the scheduled follow-up will be compared between the two groups. Follow-up time will be censored at the last available assessment in patients who will be lost to follow-up without having an event. Time from randomization to event will be summarized by Kaplan-Meier curves, and compared with the log rank test. Hazard ratios (HRs) with 95% CIs will be calculated with Cox's regression to estimate size of the treatment effect. The proportional hazards assumption will be tested formally with analysis of Schoenfeld residuals. All analyses will be performed with STATA.

Sample Size And Power It is planed to enroll 250 subjects. Based on the magnitude of effect and variation observed in our pilot clinical experience, it is projected that a sample size of 250 subjects will achieve a power of 0.80. It has been reported an Odds Ratio (OR) of 0.2 over 5 years, starting from the third and fourth decades of life, with absolute rates of 22% in mood disorder patients versus 5% in non-mood disorder controls. The mean age was 68. Based on these findings, an estimated Hazard Ratio (HR) of 0.7 for our overall sample of 250 subjects is expected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-70.
2. DSM-5 diagnosis of major depressive disorder or bipolar disorder (types I or II), current or lifetime.
3. Prior to participation in this study, each subject must sign an informed consent.

Exclusion Criteria:

1. Current mood treatment with lithium.
2. Alcohol dependency within the past month.
3. Current serious unstable medical conditions or history of medical illness that would contraindicate a trial of lithium.
4. Current or past severe kidney disease or baseline creatinine > 1.5 mg/dl.
5. Active suicidal ideation with plan and intent (Columbia Suicide Severity Rating Scale Screen Version (C-SSRS Screen) > 3 points).
6. Current or past severe thyroid disease or baseline TSH >5.0 uUI/dl.
7. Current diagnosis of dementia of any kind.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of MCI | Five years follow-up
  Incidence of Mild Cognitive Impairment (MCI) on a yearly basis from year one until the end of the study (year five). This primary outcome will be defined as change from patients initially with a Clinical Dementia Rating Scale (CDR) score of 0 to 0.5 (MCI).
  The Clinical Dementia Rating Scale is a numerical scale used to quantify the severity of symptoms of dementia. It is used for assessing six cognitive and functional domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The CDR scale helps in categorizing the stages of dementia from no dementia (CDR 0) to severe dementia (CDR 3), providing a standardized measure for the severity of dementia.
  The primary analysis will employ a Cox regression model to analyze the time to first clinical diagnosis of MCI.

SECONDARY OUTCOMES:
Clinical predictors of lithium response | Five years follow-up
  Sheehan Disability Scale (SDS): is a self-administered psychological assessment tool that measures functional impairment in three inter-related domains: work/school, social, and family life. Developed by Dr. David Sheehan, the SDS is commonly used to evaluate the extent to which mental health symptoms disrupt daily functions and responsibilities.
  It has five items with a Likert scale from 0 (not at all) to 10 (extremely). Total score 0: lack of disability Total score 1-3: mild disability Total score 4-6: moderate disability Total score 7-10: extreme disability
Clinical predictors of lithium response | Five years follow-up
  Columbia Suicide Severity Rating Scale (C-SSRS): A tool used for the assessment of suicidal ideation and behavior. It is designed to evaluate the severity of suicidal ideation and the presence of suicidal behavior in individuals. The scale has been widely adopted in clinical and research settings due to its sensitivity in identifying varying degrees of suicidality and its ability to support timely interventions.
  It has six self reported YES/NO questions addressing different context to determine low, moderate and high risk of suicide.
Clinical predictors of lithium response | Five years follow-up
  Patient Health Questionnaire-9 (PHQ-9): A widely used nine-item self-administered instrument for screening, diagnosing, monitoring and measuring the severity of depression. The scores range from 0 to 27, with a score of 10 or more indicative of a possible clinically significant depression. The PHQ-9 was validated in Chile.
  It consist of nine self reported items, four-point scale from 0 (never) to 3 (almost every day) each.
  Total score less than 5: absence of a depressive disorder Total score 5 to 9: no depression or sub-threshold depression Total scores of 10 to 14: spectrum of depression Total scores of 15 or greater: major depression
Clinical predictors of lithium response | Five years follow-up
  Altman Self-Rating Mania Scale (ASMS): Self-report questionnaire used to assess the presence and severity of mania symptoms. It is commonly used in both clinical and research settings to monitor manic episodes in individuals with mood disorders. The scale consists of five items scoring from 0 to 4 each, including elevated mood, increased energy, reduced need for sleep, and hyperactivity.
  Total total score 15-20: mild mania Total score 21 -28: moderate mania Total score 29-32: marked mania Total score 33 - 43: severe mania Total score ≥44: extreme mania
Clinical predictors of lithium response | Five years follow-up
  Shahin Mixed Depression Scale (SMDS): This instrument is specifically designed to measure non-DSM mixed features in depression. It was developed to address gaps in the traditional DSM-5 criteria, which may not fully capture the spectrum of mixed symptoms in depressive disorders. It consist of thirteen self-reported YES/NO questionnaire. The first part (items 1-6) evaluates psychomotor agitation, with a cut-off score ≥ 2. The second part (items 6-13) re-evaluates Koukopoulos' mixed depression diagnostic criteria (13), with a cut-off score ≥ 3.
Clinical predictors of lithium response | Five years follow-up
  Beck Anxiety Inventory (BAI): This is a self-report assessment tool designed to evaluate the presence and severity of anxiety symptoms. It is composed by 21 items with a four-point scale, that measure the presence and severity of anxiety symptoms such as nervousness, trembling, fear, and physical symptoms. It is widely used because of its robustness and validity in measuring anxiety.
  Total score: 0-7: minimal anxiety levels Total score 8-15: mild anxiety Total score 16-25: moderate anxiety Total score 25-63: severe anxiety
Clinical predictors of lithium response | Five years follow-up
  Montreal Cognitive Assessment (MoCA): Clinical twelve items screening instrument designed to detect mild cognitive impairments. It is primarily used to evaluate memory, orientation, concentration, and executive functions among other cognitive abilities. The MoCA is widely used to identify cognitive problems in patients who may be in the early stages of Alzheimer's disease or other forms of dementia. It has been validated in Chile.
  Total score 24-30: is considered normal for chilean population Total score 0-23: probably cognitive impairment
Clinical predictors of lithium response | Five years follow-up
  INECO frontal screening scale (IFS): A neuropsychological eight items test specifically designed to assess various frontal lobe functions including abstraction, mental flexibility, motor programming, working memory, and inhibitory control. The IFS is particularly useful for detecting early signs of executive dysfunction in neurological diseases such as frontotemporal dementia and Alzheimer's disease. It has been validated in Chile.
  Total score 18-30: normal executive functioning Total score 0-17: probable executive disfunction
Clinical predictors of lithium response | Five years follow-up
  Free and Cued Selective Reminding Test (FCSRT): Developed by Grober and Buschke, is an episodic memory test that specifically evaluates memory. It has a good discriminative ability to predict the development of Alzheimer's disease up to 5 years before its clinical onset among elderly subjects. Additionally, this test is minimally influenced by schooling factors, making it an ideal tool to detect Alzheimer's disease in individuals with low literacy levels. This test has shown appropriate accuracy in distinguishing mild Alzheimer's disease patients from controls in the Chilean population.
  Scores proposed to suspect very mild or incident dementia, identify MCI patients with higher risk for developing AD and for differentiating AD and non AD dementias are:
  1. Total Recall: < 40
  2. Free Recall: <17
  3. Total Delayed Recall: <14
Clinical predictors of lithium response | Five years follow-up
  EuroQol EQ-5D: This is a standardized five questions instrument for measuring an individual's self-reported health status. It encompasses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is assessed on a scale with three levels of severity: no problems, moderate problems, and severe problems. The corresponding values of 1 (normal), 2 (some problems), and 3 (severe problems) are assigned during data analysis to quantify the health status based on the patient's responses. The EQ-5D has been widely used in various clinical settings, including in the assessment of individuals with affective disorders.
Clinical predictors of lithium response | Five years follow-up
  MINI-International Neuropsychiatric Interview: A brief structured diagnostic psychiatric interview for DSM-IV and ICD-10 psychiatric disorders. It will be used for the diagnosis of:
  1. Alcohol dependency
  2. Abuse of psychoactive substances
  3. Bipolar disorder
  4. Major depressive disorders

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Instituto Psiquiátrico Dr. José Horwitz Barak, Santiago, Santiago Metropolitan
  - Psychiatric Institute Dr. José Horwitz Barak, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kessing LV, Sondergard L, Forman JL, Andersen PK. Lithium treatment and risk of dementia. Arch Gen Psychiatry. 2008 Nov;65(11):1331-5. doi: 10.1001/archpsyc.65.11.1331. PMID 18981345
- [Background] Angst J, Gamma A, Neuenschwander M, Ajdacic-Gross V, Eich D, Rossler W, Merikangas KR. Prevalence of mental disorders in the Zurich Cohort Study: a twenty year prospective study. Epidemiol Psichiatr Soc. 2005 Apr-Jun;14(2):68-76. doi: 10.1017/s1121189x00006278. PMID 16001703
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Shahin I, Bonnin CDM, Saleh E, Helmy K, Youssef UM, Vieta E. Validity of the Shahin Mixed Depression Scale: A Self-Rated Instrument Designed to Measure the Non-DSM Mixed Features in Depression. Neuropsychiatr Dis Treat. 2020 Sep 28;16:2209-2219. doi: 10.2147/NDT.S259996. eCollection 2020. PMID 33061391
- [Background] Altman EG, Hedeker D, Peterson JL, Davis JM. The Altman Self-Rating Mania Scale. Biol Psychiatry. 1997 Nov 15;42(10):948-55. doi: 10.1016/S0006-3223(96)00548-3. PMID 9359982
- [Background] Errazuriz A, Beltran R, Torres R, Passi-Solar A. The Validity and Reliability of the PHQ-9 and PHQ-2 on Screening for Major Depression in Spanish Speaking Immigrants in Chile: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Oct 27;19(21):13975. doi: 10.3390/ijerph192113975. PMID 36360856
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996 Jun;11 Suppl 3:89-95. doi: 10.1097/00004850-199606003-00015. PMID 8923116
- [Background] Rada I, Ortiz MS, Cabieses B. [Health-related quality of life in Chileans from vulnerable communes]. Gac Sanit. 2023 Sep 30;37:102328. doi: 10.1016/j.gaceta.2023.102328. eCollection 2023. Spanish. PMID 37783060
- [Background] Slachevsky A, Barraza P, Hornberger M, Munoz-Neira C, Flanagan E, Henriquez F, Bravo E, Farias M, Delgado C. Neuroanatomical Comparison of the "Word" and "Picture" Versions of the Free and Cued Selective Reminding Test in Alzheimer's Disease. J Alzheimers Dis. 2018;61(2):589-600. doi: 10.3233/JAD-160973. PMID 29226861
- [Background] Delgado C, Munoz-Neira C, Soto A, Martinez M, Henriquez F, Flores P, Slachevsky A. Comparison of the Psychometric Properties of the "Word" and "Picture" Versions of the Free and Cued Selective Reminding Test in a Spanish-Speaking Cohort of Patients with Mild Alzheimer's Disease and Cognitively Healthy Controls. Arch Clin Neuropsychol. 2016 Mar;31(2):165-75. doi: 10.1093/arclin/acv107. Epub 2016 Jan 11. PMID 26758367
- [Background] Jory JI, Bruna AA, Munoz-Neira C, Chonchol AS. Chilean version of the INECO Frontal Screening (IFS-Ch): psychometric properties and diagnostic accuracy. Dement Neuropsychol. 2013 Jan-Mar;7(1):40-47. doi: 10.1590/S1980-57642013DN70100007. PMID 29213818
- [Background] Torralva T, Roca M, Gleichgerrcht E, Lopez P, Manes F. INECO Frontal Screening (IFS): a brief, sensitive, and specific tool to assess executive functions in dementia. J Int Neuropsychol Soc. 2009 Sep;15(5):777-86. doi: 10.1017/S1355617709990415. Epub 2009 Jul 28. PMID 19635178
- [Background] Gaete M, Jorquera S, Bello-Lepe S, Mendoza YM, Veliz M, Alonso-Sanchez MF, Lira J. Standardized results of the Montreal Cognitive Assessment (MoCA) for neurocognitive screening in a Chilean population. Neurologia (Engl Ed). 2020 Nov 5:S0213-4853(20)30294-2. doi: 10.1016/j.nrl.2020.08.017. Online ahead of print. English, Spanish. PMID 33160725
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Figueroa LT, Razmillic B, Zumeata O, Aranda GN, Barton SA, Schull WJ, Young AH, Kamiya YM, Hoskins JA, Ilgren EB. Environmental lithium exposure in the north of Chile--II. Natural food sources. Biol Trace Elem Res. 2013 Jan;151(1):122-31. doi: 10.1007/s12011-012-9543-1. Epub 2012 Nov 28. PMID 23188677
- [Background] Nunes MA, Viel TA, Buck HS. Microdose lithium treatment stabilized cognitive impairment in patients with Alzheimer's disease. Curr Alzheimer Res. 2013 Jan;10(1):104-7. doi: 10.2174/1567205011310010014. PMID 22746245
- [Background] Nunes PV, Forlenza OV, Gattaz WF. Lithium and risk for Alzheimer's disease in elderly patients with bipolar disorder. Br J Psychiatry. 2007 Apr;190:359-60. doi: 10.1192/bjp.bp.106.029868. PMID 17401045
- [Background] Angst J, Gamma A, Gerber-Werder R, Zarate CA Jr, Manji HK. Does long-term medication with lithium, clozapine or antidepressants prevent or attenuate dementia in bipolar and depressed patients? Int J Psychiatry Clin Pract. 2007;11(1):2-8. doi: 10.1080/13651500600810133. PMID 24941269
- [Background] Haupt M, Bahr M, Doeppner TR. Lithium beyond psychiatric indications: the reincarnation of a new old drug. Neural Regen Res. 2021 Dec;16(12):2383-2387. doi: 10.4103/1673-5374.313015. PMID 33907010
- [Background] Singulani MP, Ferreira AFF, Figueroa PS, Cuyul-Vasquez I, Talib LL, Britto LR, Forlenza OV. Lithium and disease modification: A systematic review and meta-analysis in Alzheimer's and Parkinson's disease. Ageing Res Rev. 2024 Mar;95:102231. doi: 10.1016/j.arr.2024.102231. Epub 2024 Feb 15. PMID 38364914
- [Background] Mauer S, Vergne D, Ghaemi SN. Standard and trace-dose lithium: a systematic review of dementia prevention and other behavioral benefits. Aust N Z J Psychiatry. 2014 Sep;48(9):809-18. doi: 10.1177/0004867414536932. Epub 2014 Jun 11. PMID 24919696
- [Background] Kessing LV, Nilsson FM. Increased risk of developing dementia in patients with major affective disorders compared to patients with other medical illnesses. J Affect Disord. 2003 Feb;73(3):261-9. doi: 10.1016/s0165-0327(02)00004-6. PMID 12547295
- [Background] Forlenza OV, Diniz BS, Radanovic M, Santos FS, Talib LL, Gattaz WF. Disease-modifying properties of long-term lithium treatment for amnestic mild cognitive impairment: randomised controlled trial. Br J Psychiatry. 2011 May;198(5):351-6. doi: 10.1192/bjp.bp.110.080044. PMID 21525519
- [Background] Forlenza OV, De-Paula VJ, Diniz BS. Neuroprotective effects of lithium: implications for the treatment of Alzheimer's disease and related neurodegenerative disorders. ACS Chem Neurosci. 2014 Jun 18;5(6):443-50. doi: 10.1021/cn5000309. Epub 2014 May 6. PMID 24766396
- [Background] Pfennig A, Littmann E, Bauer M. Neurocognitive impairment and dementia in mood disorders. J Neuropsychiatry Clin Neurosci. 2007 Fall;19(4):373-82. doi: 10.1176/jnp.2007.19.4.373. PMID 18070839
- [Background] Wu KY, Chang CM, Liang HY, Wu CS, Chia-Hsuan Wu E, Chen CH, Chau YL, Tsai HJ. Increased risk of developing dementia in patients with bipolar disorder: a nested matched case-control study. Bipolar Disord. 2013 Nov;15(7):787-94. doi: 10.1111/bdi.12116. Epub 2013 Aug 31. PMID 23992521
- [Background] Velosa J, Delgado A, Finger E, Berk M, Kapczinski F, de Azevedo Cardoso T. Risk of dementia in bipolar disorder and the interplay of lithium: a systematic review and meta-analyses. Acta Psychiatr Scand. 2020 Jun;141(6):510-521. doi: 10.1111/acps.13153. Epub 2020 Feb 11. PMID 31954065
- [Background] Ownby RL, Crocco E, Acevedo A, John V, Loewenstein D. Depression and risk for Alzheimer disease: systematic review, meta-analysis, and metaregression analysis. Arch Gen Psychiatry. 2006 May;63(5):530-8. doi: 10.1001/archpsyc.63.5.530. PMID 16651510
- [Background] Diniz BS, Teixeira AL, Cao F, Gildengers A, Soares JC, Butters MA, Reynolds CF 3rd. History of Bipolar Disorder and the Risk of Dementia: A Systematic Review and Meta-Analysis. Am J Geriatr Psychiatry. 2017 Apr;25(4):357-362. doi: 10.1016/j.jagp.2016.11.014. Epub 2017 Jan 4. PMID 28161155
- [Background] da Silva J, Goncalves-Pereira M, Xavier M, Mukaetova-Ladinska EB. Affective disorders and risk of developing dementia: systematic review. Br J Psychiatry. 2013 Mar;202(3):177-86. doi: 10.1192/bjp.bp.111.101931. PMID 23457181
- [Background] Chen MH, Li CT, Tsai CF, Lin WC, Chang WH, Chen TJ, Pan TL, Su TP, Bai YM. Risk of subsequent dementia among patients with bipolar disorder or major depression: a nationwide longitudinal study in Taiwan. J Am Med Dir Assoc. 2015 Jun 1;16(6):504-8. doi: 10.1016/j.jamda.2015.01.084. Epub 2015 Feb 27. PMID 25737262
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Petersen RC. Mild Cognitive Impairment. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):404-18. doi: 10.1212/CON.0000000000000313. PMID 27042901
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Gillis C, Mirzaei F, Potashman M, Ikram MA, Maserejian N. The incidence of mild cognitive impairment: A systematic review and data synthesis. Alzheimers Dement (Amst). 2019 Mar 8;11:248-256. doi: 10.1016/j.dadm.2019.01.004. eCollection 2019 Dec. PMID 30911599
- [Background] Vicente B, Kohn R, Rioseco P, Saldivia S, Levav I, Torres S. Lifetime and 12-month prevalence of DSM-III-R disorders in the Chile psychiatric prevalence study. Am J Psychiatry. 2006 Aug;163(8):1362-70. doi: 10.1176/ajp.2006.163.8.1362. PMID 16877648
- [Background] Kessler RC, Akiskal HS, Ames M, Birnbaum H, Greenberg P, Hirschfeld RM, Jin R, Merikangas KR, Simon GE, Wang PS. Prevalence and effects of mood disorders on work performance in a nationally representative sample of U.S. workers. Am J Psychiatry. 2006 Sep;163(9):1561-8. doi: 10.1176/ajp.2006.163.9.1561. PMID 16946181